CLINICAL TRIAL: NCT00710112
Title: Genetic Variants and Susceptibility to Diseases of Prematurity in Very Low Birth-Weight Infants
Acronym: CLD
Status: Recruiting | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, G. Ganesh Konduri, Chief, Division of Neonatology; Professor, Medical College of Wisconsin
Other Study IDs: PRO44242
Record Dates: First submitted 2008-06-19; First posted 2008-07-04 (Estimated); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Chronic Lung Disease
Keywords: CLD; VLBW infants; Toll like Receptors; Biomarkers
MeSH Terms: interventions — Toll-Like Receptors; Biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- VLBW: infants less than 1500 grams at birth
  Interventions: Genetic: gene variations

INTERVENTIONS:
Genetic: gene variations — comparing variations in genes in infants who develop chronic lung disease and other diseases of prematurity and those who do not.
  Other Names: toll like receptors, biomarkers

SUMMARY:
The purpose of this study is to determine if sequence variations in genes involved in the development and function of vulnerable organs increases susceptibility to chronic lung disease (CLD) and other diseases affecting premature infants, such as necrotizing enterocolitis (NEC), sepsis, patent ductus arteriosus (PDA) and intraventricular hemorrhage (IVH). The study will also determine whether measurement of certain biomarkers in serum will identify infants who will develop these complications of prematurity. Previous studies from this institution and others have identified genetic variants in some genes, such as toll like receptor genes are associated with higher risk of CLD or NEC. The interaction of these variants with other gene variants that can influence the risk of these diseases remains unclear.

DETAILED DESCRIPTION:
Chronic lung disease of prematurity (CLD) is diagnosed in 30-40% of very low birth weight (VLBW) infants (<1500gms) and remains a leading cause of mortality and long-term morbidity in this population. Other diseases such as necrotizing enterocolitis (NEC), sepsis, patent ductus arteriosus (PDA), and intraventricular hemorrhage (IVH) also contribute to mortality and morbidity in this population. A central tenet in the pathogenesis of NEC, CLD and sepsis is the failure of host genome-regulated immune defenses to surmount the challenges posed by microbial pathogens in the presence of risk-factors that induce intestinal, pulmonary and systemic injury, respectively. Toll like receptors (TLRs) are pathogen recognition receptors which serve as the recognition and effector arm of the innate immune system. Since the premature infant is predominantly dependent on the innate immune system for host defense our hypothesis is that hypomorphic genetic variations in TLRs will increase susceptibility to diseases of prematurity such as CLD and sepsis.The increased risk of inflammation, decreased potential for repair and growth of lung may be reflected in the levels of biomarkers, such as, cytokines, micro-RNAs (miRNA) or peptides that are secreted into biological fluids, like blood and tracheal aspirates. It is likely that the genetic variants that increase the risk of inflammation or decreased repair and growth will be also associated with altered levels of these biomarkers. Measurement of the biomarkers and genetic variants together can increase the precision of the early predictors of these complications of prematurity. Measurement of biomarkers in biological fluids can be done with a shorter turnaround time than gene sequencing at the present time. Biomarkers can also provide longitudinal changes in the severity of disease and response to therapy. Newer multiplex assays make it feasible to measure the levels of biomarkers in very small quantities of biological fluids. These complementary strengths make gene sequencing and biomarker detection ideal 1-2 approach for the early identification and disease progression evaluation in premature infants. Our hypothesis will be tested in VLBW infants in four specific aims: (1) To determine whether the presence of previously described single nucleotide polymorphisms (SNPs) in TLR4 (Asp299Gly, Thr399Ile) TLR2 (Arg753Gln) and TLR5 (Arg392STOP) genes is associated with an increased risk of CLD ; (2) to detect by DNA sequencing if novel genetic variations in TLR4, TLR2, TLR9, MyD88 and other innate immune genes increases the risk of CLD or other disease in premature infants; (3) to identify by gene sequence approach whether variants in other repair and growth genes alter susceptibility to diseases affecting premature infants such as CLD,NEC or sepsis or PDA or IVH; and (4) whether alterations in cytokines, miRNA and other biomarker levels in serum from the same blood samples can provide additional predictive value in recognizing the risk of diseases of prematurity. VLBW infants who develop CLD (oxygen requirement at 36 weeks postconceptional age), NEC, sepsis, PDA, or IVH will serve as cases while VLBW infants who do not develop the diseases of interest will serve as controls. A 0.5cc sample of blood will be collected from enrolled infants via indwelling catheter or heel-stick for DNA analysis after consent is obtained. The TLR4 (Asp299Gly, Thr399Ile) TLR2 (Arg753Gln) and TLR5 (Arg392STOP) SNPs will be evaluated using a multiplex Single Base extension based technique, using commercially available primers. Novel genetic variations in these genes of interest and other variants proposed to be related to NEC will be detected using conventional Sanger or Next Generation DNA sequencing. Serum will be separated from the same blood sample obtained for DNA isolation. A second 0.5cc sample of blood will be collected for biomarker measurement. Biomarker levels in serum will be analyzed using multiplex EIA for cytokines, sequencing for miRNA profile and ELISA for peptide levels of interest (VEGF, angiopoietin-2 and Nogo-B peptide). Benefits include the possibility of development of risk-based preventive and therapeutic strategies to prevent CLD, NEC, sepsis, PDA, or IVH in this population.

ELIGIBILITY:
Inclusion Criteria:

* Infants born weighing less than 1500 grams

Exclusion Criteria:

* Infants born with congenital heart disease (other than patent ductus arteriosus)
* major congenital anomalies of the GI tract, respiratory tract, or kidneys

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Infants born weighing less than 1500 grams
Sampling Method: Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2006-06; Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
To determine if small variations in certain genes predispose infants to the development of chronic lung disease and other diseases of prematurity | participants will be followed for the duration of hospital stay, an expected average of 6 to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: G. Ganesh Konduri, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Wisconsin, Milwaukee, Wisconsin, United States